## Imperial College London



## **Consent Agreement**

Full Title of Project: The HeartHive COVID-19 Study

Name of Principal Investigator: James Ware

- 1 I confirm that I have read and understand the information about the HeartHive COVID-19 Study.
- I understand that my participation is voluntary and I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected.
- I agree to complete multiple online health surveys for this study. Information from these may be used in future medical and health-related studies which have relevant scientific and ethics approval.
- 4 I agree for information that I have provided to the Heart Hive Registry and Database to be released to the research team.
- I also agree to information provided for the purpose of this study being held by the Heart Hive Registry and Database.
- If I enrol in the HeartHive Cardiomyopathy Study (or if I have already enrolled in this study), then I agree for health information and genetic results from this to be released to the study team.
- 7 I understand that subjects enrolled in this study and residing in the United Kingdom will have information relating to their health collected from national electronic registries and NHS databases, hospitals and GP records over their lifetime and after death and I agree to this.
- 8 I agree to my information being stored at Imperial College.
- I agree to be contacted by the research team to be invited to participate in future medical and health-related studies which have relevant scientific and ethics approval. I understand that I do not have to participate in any future studies.
- 10 I understand that results from research on my medical information may be published on databases. I understand that no information that would reveal my identity will be included on these databases.
- I understand that my data may be shared with other researchers. This may include genetic information. I understand that information from my data will only be made available to researchers in a form that protects my identity.
- 12 I understand my data may be sent outside the EU, including to the USA.
- 13 I understand that my medical information will be treated confidentially.
- 14 I understand that sections of any of my medical notes may be looked at by responsible individuals from Imperial College or from regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to access my records that are relevant to this research
- 15 I agree to take part in the above study.

| Name of Subject | Date |
|-----------------|------|